CLINICAL TRIAL: NCT01221012
Title: Heat Stress and Physiological Strain of Permeable vs. Impermeable CB Protective Garment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, amit druyan, Principal Investigator, Medical Corps, Israel Defense Force
Other Study IDs: 883-2009-CLIT
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Heat Tolerance

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (5):
- men wearing Semipermeable garment
- air permeable garment type BP2
- air permeable garment type BP3
- air permeable garment type MO
- air permeable garment type BP1

SUMMARY:
Current protective clothing of any kind, especially the nuclear-biological-chemical (NBC) protective garments, amplify thermal stress because of the inherent properties of the clothing material. High insulation coefficient and low water vapor permeability of the protective cloth limit the ability of sweat to readily evaporate, which consequently result with a significant elevation of body temperature and with excessive body fluid loss (because of inefficient sweating) that might result with significant dehydration.

Combat soldiers require to perform intense physical activities under hostile environmental conditions, including in contaminated areas that need the use of protective garments. The ability to fulfill a mission derives from the soldier's professionalism and from his physiological limits. It is well established that wearing protective garments affect tolerance time (TT) and performance.

To operate in contaminated areas suitable protective garments should be worn. The inherent characteristics of the current protective garments limit, however, the effective working periods with such an ensemble, which is further aggravated in hot climate. Thus, in an attempt to increase TT and enhance work effectiveness, improved protective garments, which result with a lessened heat-stress, are under different stages of development.

The relative influence of air permeability properties, garment weight and garment construction on heat stress and physiological strain will be investigated.

The results will be quantified in terms of body temperatures, heart rate, fluid balance, subjective sensation and the maximum wear time (if necessary extrapolated).

ELIGIBILITY:
Inclusion Criteria:

* Twelve young (20-30 yr) male subjects will voluntarily participate in this study. The potential participants will be informed of the study's nature, purpose and medical risks. Their inclusion in the study requires the medical clearance by the study's physician (CRF) and after having filled out and sign an informed consent form

Exclusion Criteria:

* heart conditions, blood pressure higher than 140/90 mmHg, known diabetes or any skin illness or lesions. Also be excluded are potential participants who were ill during the 2 weeks prior to the study

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twelve young (20-30 yr) male subjects will voluntarily participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The physiological burden of different CB Protective Garments | 1 year
  The physiological burden of different CB Protective Garments will be mesured by a heat tolerance test (HTT).
  The subjects will undergo an HTT wearing different CB Protective Garments and the results which indicate physiological burden will be compared between the different garments.

SECONDARY OUTCOMES:
Rectal temperature | 1 year
  The rectal temperature will be mesured by rectal thermistore.
Skin temperature | 1 year
  The skin temperature will be mesured by skin thermistores conected to 3 different sites (chest, leg and arm).
Heart rate | 1 year
  Heart rate will be mesured by a polar watch.
Sweat rate | 1 year
  The sweat rate will be calculated in each HTT from the subject's weight before and after the test and his water balance.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Druyan, M.D, Principal Investigator — Medical Corps, Israel Defense Force
Locations (1):
- Sheba medical center, Ramat Gan, Israel